CLINICAL TRIAL: NCT01701258
Title: Early Life Stress and Depression: Molecular and Functional Imaging Approaches
Brief Title: An Investigation of Early Life Stress and Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Associate Professor of Psychiatry, Harvard Medical School, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012P002593; 5R01MH095809 (NIH)
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder (MDD); History of Childhood Sexual Abuse (CSA)
Keywords: Depression; Childhood Sexual Abuse; Dopamine; MRI; PET; ERP; Stress; Reward; Childhood trauma; Amisulpride
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Amisulpride

STUDY DESIGN:
Intervention Model Description: There were four groups of subjects: those with a history of child sexual abuse that are currently experiencing a major depressive episode, those with a history of child sexual abuse without a current or past diagnosis of major depressive disorder, those without a history of child sexual abuse that are currently experiencing a major depressive episode, and those with without a history of child sexual abuse and without a current or past diagnosis of major depressive disorder. Within each group, half of the subjects were assigned to receive the study drug (amisulpride) and half to receive a placebo for the fMRI session (session 2 or 3).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- CSA/MDD-amisulpride (Active Comparator): Subjects experiencing a current episode of major depression (MDD) with a history of child sexual abuse (CSA) are randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session.
  Interventions: Drug: Amisulpride
- CSA/MDD-placebo (Placebo Comparator): Subjects experiencing a current episode of major depression (MDD) with a history of child sexual abuse (CSA) are randomized to receive a placebo during the fMRI session.
  Interventions: Drug: Placebo
- CSA/RES-amisulpride (Active Comparator): Subjects with a history of child sexual abuse (CSA) without a current or past diagnosis of major depressive disorder (RES) are randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session.
  Interventions: Drug: Amisulpride
- CSA/RES-placebo (Placebo Comparator): Subjects with a history of child sexual abuse (CSA) without a current or past diagnosis of major depressive disorder (RES) are randomized to receive a placebo during the fMRI session.
  Interventions: Drug: Placebo
- MDD-amisulpride (Active Comparator): Subjects without a history of child sexual abuse that are currently experiencing a major depressive episode are randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session.
  Interventions: Drug: Amisulpride
- MDD-placebo (Placebo Comparator): Subjects without a history of child sexual abuse that are currently experiencing a major depressive episode are randomized to receive a placebo during the fMRI session.
  Interventions: Drug: Placebo
- Control-amisulpride (Active Comparator): Subjects without a history of child sexual abuse and without a current or past diagnosis of major depressive episode are randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session.
  Interventions: Drug: Amisulpride
- Control-placebo (Placebo Comparator): Subjects without a history of child sexual abuse and without a current or past diagnosis of major depressive episode are randomized to receive a placebo during the fMRI session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amisulpride — single low-dose pharmacological challenge, 50 mg amisulpride during the fMRI session only
  Other Names: Solian
  Arms: CSA/MDD-amisulpride; CSA/RES-amisulpride; Control-amisulpride; MDD-amisulpride
Drug: Placebo — single-dose placebo capsule during the fMRI session only
  Arms: CSA/MDD-placebo; CSA/RES-placebo; Control-placebo; MDD-placebo

SUMMARY:
The purpose of this study is to investigate brain pathways within adult females (with a history of CSA that occurred between the ages of 5-14) with and without a current diagnosis of major depressive disorder (MDD).

Hypotheses:

The CSA/MDD participants will be characterized by (1) reduced reward responsiveness and prefrontal cortex activity, but increased cortisol levels, (2) reduced dopamine activity, and (3) reduced dopamine transporter binding. The over-arching purpose of the study is to (1) identify individuals at risk for psychopathology and maladaptive behavior, (2) prevent re-victimization, and (3) develop more targeted therapeutic interventions.

DETAILED DESCRIPTION:
This study will include four sessions:

Session 1 (SCID Session) The first session takes place at the Center for Depression, Anxiety, and Stress Research (CDASR) or Neuroimaging Center (both at McLean Hospital) and involves consenting, a clinical evaluation, a series of questionnaires, and a medical assessment.

Session 2 or 3 (fMRI Session) The third session takes place at the Neuroimaging Center. Using a double-blind design, participants will be administered either amisulpride (50 mg) or placebo. Participants will complete the Monetary Incentive Delay (MID) task during functional magnetic resonance imaging (fMRI) and the Probabilistic Stimulus Selection Task (PSST) afterwards.

Session 2 or 3 (PET Session) This session takes place at Massachusetts General Hospital. 9 mCi of [11C] altropane will be injected by a trained nuclear medicine technician and positron emission tomography (PET) scanning will begin. Prior to the PET scan, a blood serum pregnancy test will be administered for females.

Session 4 (ERP Session) The fourth session takes place at the CDASR and involves an electroencephalography (EEG) recording, the Probabilistic Reward Task (PRT), and collecting saliva samples to assess cortisol levels.

ELIGIBILITY:
General Inclusion Criteria:

* Females of all ethnic origins, age between 20 and 45; right-handed (Chapman & Chapman 1987);
* Absence of any psychotropic medications for at least 2 weeks (6 weeks for fluoxetine; 6 months for neuroleptics; 2 weeks for benzodiazepines; 2 weeks for any other antidepressants);

Inclusion Criteria for Childhood Sexual Abuse/MDD (CSA/MDD) Group:

* At least one incident of contact sexual abuse1 between the ages 5-14 years;
* Current DSM-IV diagnostic criteria for MDD (as diagnosed with the use of the SCID);

Inclusion Criteria for Childhood Sexual Abuse/Resilient (CSA/RES) Group:

* At least one incident of contact sexual abuse1 between the ages 5-14 years;
* Absence of past or current DSM diagnosis, including MDD or alcohol/substance abuse;

Inclusion Criteria for Non-traumatized, MDD (MDD) Group:

* No incidents of sexual, verbal, or physical abuse (ascertained using the Traumatic Antecedents Questionnaire);
* Current DSM-IV diagnostic criteria for MDD (as diagnosed with the use of SCID);

Non-traumatized, healthy controls (controls):

* No incidents of sexual, verbal, or physical abuse (ascertained using the Traumatic Antecedents Questionnaire);
* Absence of any medical, neurological, and psychiatric illness (including alcohol/substance abuse)

Exclusion Criteria:

* Participants with suicidal ideation where study participation is deemed unsafe by the study clinician;
* Pregnant women or women of childbearing potential who are not compliant with the requirements of a urine and blood pregnancy test.
* Failure to meet MRI or PET safety requirements.
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine (hypothyroidism), neurologic or hematologic disease;
* Past/current DSM diagnosis of: OCD, ADHD, schizophrenia, schizoaffective disorder, delusional disorder, bipolar disorder, mood congruent/incongruent psychotic features, substance dependence, substance abuse within the last 12 months (with the exception of cocaine or stimulant abuse, which will lead to automatic exclusion);
* Simple phobia, social anxiety disorder and generalized anxiety disorders will be allowed only if secondary to MDD and only in the CSA/MDD and MDD groups (which will be matched for comorbidities);
* History of seizure disorder; renal insufficiency; history of adverse reactions to amisulpride;
* History of cocaine, stimulant, and other DA drug use [e.g., (meth)amphetamine), methylphenidate].

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaiser RH, Clegg R, Goer F, Pechtel P, Beltzer M, Vitaliano G, Olson DP, Teicher MH, Pizzagalli DA. Childhood stress, grown-up brain networks: corticolimbic correlates of threat-related early life stress and adult stress response. Psychol Med. 2018 May;48(7):1157-1166. doi: 10.1017/S0033291717002628. Epub 2017 Sep 25. PMID 28942738
- [Derived] Liu Y, Admon R, Mellem MS, Belleau EL, Kaiser RH, Clegg R, Beltzer M, Goer F, Vitaliano G, Ahammad P, Pizzagalli DA. Machine Learning Identifies Large-Scale Reward-Related Activity Modulated by Dopaminergic Enhancement in Major Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Feb;5(2):163-172. doi: 10.1016/j.bpsc.2019.10.002. Epub 2019 Oct 22. PMID 31784354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at McLean Hospital (Belmont, MA) between August, 2013, and June, 2017. The study was advertised using flyers, and on a number of internet bulletin boards available to the general public. Study visits were conducted in research facilities at McLean Hospital and Massachusetts General Hospital.
Pre-assignment Details: In session 1, subjects had a diagnostic interview, a physical exam, provided a blood sample, and completed surveys, to determine eligibility. Those eligible were invited to participate in the other sessions. Participants did not need to complete all sessions. The order depended on facility availability and convenience for participants.
Groups:
- All Participants: All participants that went through the assessment (session 1) regardless if they were eligible or ineligible.
- Control Group: Subjects without a history of child sexual abuse and without a current or past diagnosis of major depressive episode.
- Control-amisulpride (fMRI Session): After the screening visit, eligible control subjects without a history of child sexual abuse and without a current or past diagnosis of major depression were invited to participate in the fMRI session. Those that were interested were randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible baseline control participants did not complete this session.
- Control-placebo (fMRI Session): After the screening visit, eligible control subjects without a history of child sexual abuse and without a current or past diagnosis of major depression were invited to participate in the fMRI session. Those that were interested were randomized to receive a placebo during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible baseline control participants did not complete this session.
- MDD Group: Subjects without a history of child sexual abuse that are currently experiencing a major depressive episode .
- MDD-amisulpride (fMRI Session): After the screening visit, eligible subjects without a history of child sexual abuse that are currently experiencing a major depressive episode were invited to participate in the fMRI session. Those that were interested in participating, were randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible MDD baseline participants did not complete this session.
- MDD-placebo (fMRI Session): After the screening visit, eligible subjects without a history of child sexual abuse that are currently experiencing a major depressive episode were invited to participate in the fMRI session. Those that were interested in participating, were randomized to receive a placebo during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible MDD baseline participants did not complete this session.
- CSA/RES: Subjects with a history of CSA but no psychopathology ("resilient group"; CSA/RES).
- CSA/RES-amisulpride (fMRI Session): After the screening visit, eligible subjects with a history of CSA but no psychopathology ("resilient group"; CSA/RES) were invited to participate in the fMRI session. Those that were interested in participating, were randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session.This arm is specific to those that competed the fMRI session. Many eligible CSA/RES baseline participants did not complete this session.
- CSA/RES-placebo (fMRI Session): After the screening visit, eligible subjects with a history of CSA but no psychopathology ("resilient group"; CSA/RES) were invited to participate in the fMRI session. Those that were interested in participating, were randomized to receive a placebo during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible CSA/RES baseline participants did not complete this session.
- CSA/MDD Group: Subjects experiencing a current episode of major depression (MDD) with a history of child sexual abuse (CSA).
- CSA/MDD-amisulpride (fMRI Session): After the screening visit, eligible subjects with a current episode of major depression (MDD) with a history of child sexual abuse (CSA) were invited to participate in the fMRI session. Those that were interested in participating, were randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session.This arm is specific to those that competed the fMRI session. Many eligible CSA/MDD baseline participants did not complete this session.
- CSA/MDD-placebo (fMRI Session): After the screening visit, eligible subjects with a current episode of major depression (MDD) with a history of child sexual abuse (CSA) were invited to participate in the fMRI session. Those that were interested in participating, were randomized to receive a placebo. This arm is specific to those that competed the fMRI session.
  Many eligible CSA/MDD baseline participants did not complete this session.
Period: Assessment and Scheduling
Arm/Group | All Participants | Control Group | Control-amisulpride (fMRI Session) | Control-placebo (fMRI Session) | MDD Group | MDD-amisulpride (fMRI Session) | MDD-placebo (fMRI Session) | CSA/RES | CSA/RES-amisulpride (fMRI Session) | CSA/RES-placebo (fMRI Session) | CSA/MDD Group | CSA/MDD-amisulpride (fMRI Session) | CSA/MDD-placebo (fMRI Session)
Started (153 individuals were enrolled in the study. 96 were eligible after the screening visit.) | 153 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eligible After Screening Visit (96 participants were eligible after the screening visit. These were our baseline participants.) | 96 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Returned for Drug+fMRI (Session 2) (68 out of the 96 eligible participants completed the MRI.) | 68 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Returned for PET (Session 3) (73 /96 eligible completed the PET. They didn't need to complete the the MRI to complete the PET.) | 73 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Returned for EEG (Session 4) (66/96 completed the EEG. Participants did at least two sessions after the screening visit.) | 66 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Participants completed the study if they completed the screening session and two imaging sessions.) | 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 83 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Found to be Ineligible | 57 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Terminated | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Drug+fMRI (Session 2)
Arm/Group | All Participants | Control Group | Control-amisulpride (fMRI Session) | Control-placebo (fMRI Session) | MDD Group | MDD-amisulpride (fMRI Session) | MDD-placebo (fMRI Session) | CSA/RES | CSA/RES-amisulpride (fMRI Session) | CSA/RES-placebo (fMRI Session) | CSA/MDD Group | CSA/MDD-amisulpride (fMRI Session) | CSA/MDD-placebo (fMRI Session)
Started (Eligible participants after the screening session were invited to participate in this session.) | 0 | 0 | 11 | 11 | 0 | 9 | 8 | 0 | 6 | 6 | 0 | 10 | 7
Received Drug Challenge (Not all participants that were eligible completed the MRI.) | 0 | 0 | 11 | 11 | 0 | 9 | 8 | 0 | 6 | 6 | 0 | 10 | 7
Completed | 0 | 0 | 11 | 11 | 0 | 9 | 8 | 0 | 6 | 6 | 0 | 10 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PET (Session 3)
Arm/Group | All Participants | Control Group | Control-amisulpride (fMRI Session) | Control-placebo (fMRI Session) | MDD Group | MDD-amisulpride (fMRI Session) | MDD-placebo (fMRI Session) | CSA/RES | CSA/RES-amisulpride (fMRI Session) | CSA/RES-placebo (fMRI Session) | CSA/MDD Group | CSA/MDD-amisulpride (fMRI Session) | CSA/MDD-placebo (fMRI Session)
Started (Not all participants that were eligible or completed the MRI completed the PET.) | 0 | 20 | 0 | 0 | 16 | 0 | 0 | 19 | 0 | 0 | 18 | 0 | 0
Completed | 0 | 20 | 0 | 0 | 16 | 0 | 0 | 19 | 0 | 0 | 18 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: EEG (Session 4)
Arm/Group | All Participants | Control Group | Control-amisulpride (fMRI Session) | Control-placebo (fMRI Session) | MDD Group | MDD-amisulpride (fMRI Session) | MDD-placebo (fMRI Session) | CSA/RES | CSA/RES-amisulpride (fMRI Session) | CSA/RES-placebo (fMRI Session) | CSA/MDD Group | CSA/MDD-amisulpride (fMRI Session) | CSA/MDD-placebo (fMRI Session)
Started (Not all participants that were eligible or completed the MRI/PET completed the EEG.) | 0 | 19 | 0 | 0 | 14 | 0 | 0 | 16 | 0 | 0 | 17 | 0 | 0
Completed | 0 | 19 | 0 | 0 | 14 | 0 | 0 | 16 | 0 | 0 | 17 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Our baseline population are the 96 individuals that were eligible for the study after the screening visit. Not all participants that were eligible after the screening visit went on to participate in the other study sessions. Baseline data were collected for all eligible participants in each cohort during the assessment and scheduling period.
Groups:
- MDD Group: Subjects without a history of child sexual abuse that are currently experiencing a major depressive episode are randomized to receive a single low-dose pharmacological challenge.
- CSA/RES Group: Subjects with a history of CSA but no psychopathology ("resilient group"; CSA/RES).
- CSA/MDD Group: Subjects experiencing a current episode of major depression (MDD) with a history of child sexual abuse (CSA) are randomized to receive a single low-dose pharmacological challenge.
- Total: Total of all reporting groups
Arm/Group | Control Group | MDD Group | CSA/RES Group | CSA/MDD Group | Total
Number analyzed (Participants) | 26 | 17 | 24 | 29 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 17 | 24 | 29 | 96
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.44 (6.64) | 27.19 (5.99) | 25.61 (4.94) | 29.95 (6.91) | 26.63 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 17 | 24 | 29 | 96
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 2 | 0 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 9 | 5 | 21
  White | 18 | 11 | 14 | 13 | 56
  More than one race | 2 | 0 | 1 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 17 | 24 | 29 | 96
BDI II [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Beck Depression Inventory-II (BDI-II). Measures the presence and severity of 21 depressive symptoms during the past two weeks, on a scale from 0 (none, or no change) to 3 (persistent, or worsening).Range: 0 to 63. Higher scores indicate greater symptom severity. Clinical categories for total score: 0-14: absent; 14-19: mild; 20-28: moderate; 29-63: severe.
  units on a scale | 1.68 (2.79) | 27.23 (8.44) | 3.83 (5.77) | 31.49 (9.05) | 15.95 (15.14)
MASQ total [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Mood and Anxiety Symptom Questionnaire (MASQ), short form. Measures the severity of anxiety and depressive symptoms.62 items, rating of how much you have experienced certain feelings, emotions, or behaviors in the past week; item responses are on a 5-point scale from 1 (not at all) to 5 (extremely).
  Range: 62-310; higher scores indicates more severe symptoms.
  units on a scale | 93.04 (16.27) | 167.86 (22.60) | 101.82 (26.19) | 180.57 (21.89) | 135.42 (44.65)

OUTCOME MEASURES:

1. Primary Outcome: Dopamine Active Transporter Binding Potential
Description: Utilizing 11C-altropane during positron emission tomography (PET) scanning allows us to measure dopamine active transporter (DAT) binding potential.
  Our outcome measure is Nondisplacable Binding Potential (BPND). BPND refers to the ratio at equilibrium of specifically bound radioligand to that of nondisplaceable radioligand in tissue.
  *Higher BPND scores indicate greater binding potential
Time Frame: 1 hour PET scan (Session 3)
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Control Group | MDD Group | CSA/RES Group | CSA/MDD Group
Number analyzed (Participants) | 20 | 16 | 19 | 18
Ratio
  Caudate | 3.191 (0.124) | 3.161 (0.139) | 3.175 (0.130) | 3.216 (0.136)
  Putamen | 3.361 (0.120) | 3.359 (0.134) | 3.241 (0.125) | 3.318 (0.131)
  Accumbens | 2.159 (0.109) | 2.103 (0.122) | 2.103 (0.122) | 2.149 (0.119)

2. Primary Outcome: The Effects of CSA and Diagnosis on PRT Performance Under Acute Stress
Description: The participant's performance on the Probabilistic Reward Task (PRT) was assessed both before and after an acute stressor. The PRT is a behavioral task that measures an individual's ability to learn from rewarding stimuli and incorporate this learning into their response style (response bias). The acute stressor was the Maastricht Acute Stress Test (MAST). The score obtained is a ratio of the number of times participants correctly choose the high reward stimuli versus the low rewarding stimuli. Response bias scores range between -1 and +1. Higher response bias scores indicate a stronger response bias toward high reward stimuli. A negative response bias indicates a stronger bias toward low reward stimuli.
Time Frame: 3 hour EEG Session (Session 4)
Measure: Mean (Standard Deviation); unit: Ratio (Response Bias Score)
Arm/Group | Control Group | MDD Group | CSA/RES Group | CSA/MDD Group
Number analyzed (Participants) | 19 | 14 | 16 | 17
Ratio (Response Bias Score)
  PRT Block1: Before MAST | 0.028 (0.035) | 0.117 (0.045) | 0.092 (0.043) | 0.167 (0.070)
  PRT Block2: Before MAST | 0.124 (0.046) | 0.155 (0.048) | 0.130 (0.082) | 0.168 (0.102)
  PRT Block1: After MAST | 0.128 (0.026) | 0.078 (0.055) | 0.079 (0.042) | 0.048 (0.042)
  PRT Block2: After MAST | 0.245 (0.041) | 0.128 (0.035) | 0.143 (0.052) | 0.127 (0.050)

3. Primary Outcome: The Effect of Major Depressive Disorder and Childhood Abuse History on a Reward-related EEG Component (Reward Positivity Component) While Under Stress
Description: EEG was recorded during the probabilistic reward task (the PRT task). Participants completed the Probabilistic Reward Task (PRT) twice throughout the experiment, once before stress and once after stress. The stressor was the Maastricht Acute Stress Test (MAST). This statistic shows the effect that childhood sexual abuse (CSA) and diagnosis had on a reward-related positivity EEG component recorded during the PRT, before and after stress.
  * Higher reward positivity amplitudes indicate a stronger neural response to reward and lower amplitudes indicate a lower neural response to rewards.
Time Frame: 3 hour EEG Session (Session 4)
Measure: Mean (Standard Error); unit: amplitude (microvolts)
Arm/Group | Control Group | MDD Group | CSA/RES Group | CSA/MDD Group
Number analyzed (Participants) | 19 | 14 | 16 | 17
amplitude (microvolts)
  Pre MAST | 2.71 (0.86) | 4.75 (1.15) | 2.16 (0.92) | 4.15 (0.96)
  Post MAST | 2.06 (0.91) | 4.99 (1.22) | 2.30 (0.98) | 3.90 (1.01)

4. Primary Outcome: Cortisol Output in Response to a Stress Manipulation
Description: This statistic shows the impact of the stress manipulation on the participant's salivary cortisol output. Saliva samples were collected at 5 distinct time points throughout the study session. The first saliva sample (Cort 1) was collected when the participant began the eeg session. The second (Cort 2)was taken at the end of the acute stressor. The third (Cort 3) was taken approximately fifteen minutes after the second. The fourth (Cort 4) was taken approximately ten minutes after the third. The fifth (Cort 5) was taken approximately 40 minutes after the fourth.
Time Frame: 3 hour EEG Session (Session 4)
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Control Group | MDD Group | CSA/RES Group | CSA/MDD Group
Number analyzed (Participants) | 19 | 14 | 16 | 17
ng/ml
  Cort1 | 9.80 (1.27) | 12.53 (2.11) | 10.15 (2.27) | 14.19 (1.51)
  Cort2 | 9.11 (2.44) | 12.28 (1.70) | 9.51 (1.89) | 8.63 (0.95)
  Cort3 | 15.55 (4.91) | 15.23 (1.65) | 10.75 (2.19) | 14.31 (2.15)
  Cort4 | 12.89 (4.07) | 16.30 (3.24) | 8.99 (1.75) | 14.22 (2.74)
  Cort5 | 7.07 (1.80) | 10.34 (1.15) | 7.41 (1.36) | 11.01 (2.15)

5. Primary Outcome: Effects on Major Depressive Disorder and Childhood Sexual Abuse History on Striatal Activity in Response to Neutral and Reward Cues
Description: This statistic shows the influence of major depressive disorder and childhood sexual abuse history on the strength of striatal activation (caudate, putamen, accumbens) in response to neutral and reward cues during the monetary incentive delay task (MID).
  Striatal activation is measured using a statistic called a beta weight. A beta weight is a standardized regression coefficient. Higher beta weights mean greater striatal activation and lower beta weights mean less striatal activation. A negative beta weight would indicate a deactivation.
Time Frame: 3 hour Drug & fMRI Session (Session 2)
Measure: Mean (Standard Error); unit: beta weight (slope)
Arm/Group | CSA/MDD-amisulpride | CSA/MDD-placebo | CSA/RES-amisulpride | CSA/RES-placebo | MDD-amisulpride | MDD-placebo | Control-amisulpride | Control-placebo
Number analyzed (Participants) | 10 | 7 | 6 | 6 | 9 | 8 | 11 | 11
beta weight (slope)
  Caudate Response to Reward Cues | .514 (.199) | .054 (.238) | .511 (.257) | .079 (.257) | .403 (.209) | .608 (.222) | .200 (.189) | .468 (.189)
  Caudate Response to Neutral Cues | .254 (.161) | -.243 (.192) | .050 (.208) | -.370 (.208) | .047 (.170) | .156 (.180) | .222 (.154) | .185 (.154)
  Putamen Response to Reward Cues | .550 (.175) | .468 (.209) | .745 (.226) | .419 (.226) | .698 (.185) | .814 (.196) | .608 (.162) | .663 (.167)
  Putamen Response to Neutral Cues | .550 (.175) | .357 (.168) | .493 (.181) | .240 (.181) | .384 (.148) | .621 (.157) | .455 (.134) | .518 (.134)
  Accumbens Response to Reward Cues | .692 (.206) | .255 (.247) | .679 (.267) | .310 (.267) | .351 (.218) | .428 (.231) | .401 (.197) | .480 (.197)
  Accumbens Response to Neutral Cues | .385 (.173) | .040 (.207) | -.123 (.224) | -.381 (.224) | -.111 (.183) | .140 (.194) | .016 (.165) | .120 (.165)

6. Primary Outcome: Effects on Major Depressive Disorder and Childhood Sexual Abuse History on Striatal Activity in Response to Neutral and Reward Feedback
Description: This statistic shows the influence of major depressive disorder and childhood sexual abuse history on the strength of striatal activation (caudate, putamen, accumbens) in response to neutral and reward feedback during the monetary incentive delay task (MID).
  Striatal activation is measured using a statistic called a beta weight. A beta weight is a standardized regression coefficient. Higher beta weights mean greater striatal activation and lower beta weights mean less striatal activation. A negative beta weight would indicate a deactivation.
Time Frame: 3 hour Session 2 (fMRI session)
Measure: Mean (Standard Error); unit: beta weight (slope)
Arm/Group | CSA/MDD-amisulpride | CSA/MDD-placebo | CSA/RES-amisulpride | CSA/RES-placebo | MDD-amisulpride | MDD-placebo | Control-amisulpride | Control-placebo
Number analyzed (Participants) | 10 | 7 | 6 | 6 | 9 | 8 | 11 | 11
beta weight (slope)
  Caudate Response to Reward Feedback | -.101 (.329) | .040 (.393) | -.197 (.425) | -.905 (.425) | -.819 (.347) | -.773 (.368) | -.613 (.314) | -.273 (.314)
  Caudate Response to Neutral Feedback | -.233 (.314) | -.608 (.376) | -.501 (.406) | -.959 (.406) | -.865 (.331) | -.733 (.352) | -.793 (.300) | -.105 (.300)
  Putamen Response to Reward Feedback | -.018 (.217) | .063 (.260) | -.087 (.281) | -.304 (.281) | -.031 (.229) | -.357 (.243) | -.533 (.207) | -.131 (.207)
  Putamen Response to Neutral Feedback | -.021 (.201) | -.418 (.240) | -.142 (.260) | -.276 (.260) | -.229 (.221) | -.108 (.225) | -.375 (.192) | .164 (.192)
  Accumbens Response to Reward Feedback | -.158 (.421) | .839 (.503) | -.046 (.544) | -.713 (.544) | -.554 (.444) | -.215 (.471) | .074 (.401) | .069 (.401)
  Accumbens Response to Neutral Feedback | .010 (.308) | -.332 (.368) | -.079 (.398) | -.819 (.398) | -.456 (.325) | -.039 (.345) | -.503 (.294) | .109 (.294)

7. Primary Outcome: The Effect of Diagnosis on Cortisol Reactivity
Description: This is a measure of area under the curve in relation to ground, a measure of total cortisol output, in response to acute stress. The acute stressor was the Maastricht Acute Stress Test (MAST). The area under the curve includes all 5 cortisol measures, with one measure before the stressor and the other four measures collected after the stressor. Given that the cortisol data were positively skewed, the cortisol measures were normalized via a log transformation prior to calculating the area under the curve.
  Area under the curve with respect to ground (AUCG) is calculated AUC_g=(((cort2_log + cort1_log) * cort_t1_time) / 2)+(((cort3_log+cort2_log)*cort_t2_time)/2)+(((cort4_log+cort3_log)*cort_t3_time)/2)+(((cort5_log+cort4_log)*cort_t4_time)/2). Cort_logs are the log transformed cortisol output data (ng/ml) and the cort_times are the time spans in between each cortisol assessment.
Time Frame: 3 hour EEG Session (Session 4)
Measure: Mean (Standard Error); unit: [log (ng/ml)]*min
Arm/Group | Control Group | MDD Group | CSA/RES Group | CSA/MDD Group
Number analyzed (Participants) | 19 | 14 | 16 | 17
[log (ng/ml)]*min | 156.58 (10.72) | 186.78 (12.20) | 152.13 (12.20) | 179.16 (11.25)

ADVERSE EVENTS:
Time Frame: 3 years, 10 months
Groups:
- All Baseline Participants: Participants that were eligible for the study after the screening visit (session 1). These participants were invited to participate in the other study sessions.
- Control Group: Control subjects without a history of child sexual abuse and without a current or past diagnosis of major depressive episode. These participants were eligible after the screening session (session 1) and are accounted for regardless if they completed other study sessions.
- Control-amisulpride (fMRI Session): After the screening visit, eligible control subjects without a history of child sexual abuse and without a current or past diagnosis of major depression were invited to participate in the fMRI session. Those that were interested, were randomized to receive a single low-dose pharmacological challenge, 50mg amisulpride tablet during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible baseline control participants did not complete this session.
- Control-placebo (fMRI Session): After the screening visit, eligible control subjects without a history of child sexual abuse and without a current or past diagnosis of major depression were invited to participate in the fMRI session. Those that were interested, were randomized to receive a placebo during the fMRI session. This arm is specific to those that competed the fMRI session. Many eligible baseline control participants did not complete this session.
- MDD Group: Subjects without a history of child sexual abuse that are currently experiencing a major depressive episode. These participants were eligible after the screening session (session 1) and are accounted for regardless if they completed other study sessions.
- CSA/RES: Subjects with a history of CSA but no psychopathology ("resilient group"; CSA/RES). These participants were eligible after the screening session (session 1) and are accounted for regardless if they completed other study sessions.
- CSA/MDD Group: Subjects experiencing a current episode of major depression (MDD) with a history of child sexual abuse (CSA). These participants were eligible after the screening session (session 1) and are accounted for regardless if they completed other study sessions.
Arm/Group | All Participants | All Baseline Participants | Control Group | Control-amisulpride (fMRI Session) | Control-placebo (fMRI Session) | MDD Group | MDD-amisulpride (fMRI Session) | MDD-placebo (fMRI Session) | CSA/RES | CSA/RES-amisulpride (fMRI Session) | CSA/RES-placebo (fMRI Session) | CSA/MDD Group | CSA/MDD-amisulpride (fMRI Session) | CSA/MDD-placebo (fMRI Session)
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/96 | 0/26 | 0/11 | 0/11 | 0/17 | 0/9 | 0/8 | 0/24 | 0/6 | 0/6 | 0/29 | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/96 | 0/26 | 0/11 | 0/11 | 0/17 | 0/9 | 0/8 | 0/24 | 0/6 | 0/6 | 0/29 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/153 | 0/96 | 0/26 | 0/11 | 0/11 | 0/17 | 0/9 | 0/8 | 0/24 | 0/6 | 0/6 | 0/29 | 0/10 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=153) | All Baseline Participants (N=96) | Control Group (N=26) | Control-amisulpride (fMRI Session) (N=11) | Control-placebo (fMRI Session) (N=11) | MDD Group (N=17) | MDD-amisulpride (fMRI Session) (N=9) | MDD-placebo (fMRI Session) (N=8) | CSA/RES (N=24) | CSA/RES-amisulpride (fMRI Session) (N=6) | CSA/RES-placebo (fMRI Session) (N=6) | CSA/MDD Group (N=29) | CSA/MDD-amisulpride (fMRI Session) (N=10) | CSA/MDD-placebo (fMRI Session) (N=7)
Other Adverse Events (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The choice of a 50-mg dose of amisulpride was based on animal work showing low doses potentiate striatal dopamine release, have strong hedonic effects, and increase the incentive value of environmental cues. Higher doses may have different results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT01701258/Prot_SAP_000.pdf